CLINICAL TRIAL: NCT07012161
Title: Effect of Vitamin D3 Supplementation on Symptomatic Uterine Fibroid in Women With Vitamin D Deficiency
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Nahida Akter (Other)
Responsible Party: Sponsor-Investigator, Nahida Akter, Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Organization: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5256
Record Dates: First submitted 2025-04-04; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-05

CONDITIONS: Symptomatic Uterine Fibroid
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pt with uterine fibroid (Experimental): Study subjects will be selected according to inclusion and exclusion criteria, consents will be taken in informed written consent form, and then preceded as follow- 39 diagnosed women with uterine fibroid aged 18 to 50 years experiencing heavy menstrual bleeding will be purposively selected upon meeting the selection criteria Demographic information, medical history, clinical examination findings, and other relevant clinical data will be gathered through interviews Baseline Assessments: menstrual blood loss, hemoglobin concentration and ultrasound parameters (uterine volume, fibroid characteristics) Participants received 25(OH) Vitamin D3 orally
  Interventions: Drug: Colecalciferol (Vitamin D3) 50000 UI

INTERVENTIONS:
Drug: Colecalciferol (Vitamin D3) 50000 UI — Participants will received vit d upto 6 months

SUMMARY:
39 women with symptomatic uterine fibroid with serum vitamin D deficiency will receive vitamin D3 supplementation for 6 month.then symptoms and size of fibroid will be re evaluated..

DETAILED DESCRIPTION:
Effects of vitamin D supplimentation on symptomatic uterine fibroid will be checked

ELIGIBILITY:
Inclusion Criteria:

.Women aged between 18-50 not currently pregnant, lactating, or planning to conceive during the study period.

* Women with a confirmed diagnosis of uterine fibroids (leiomyoma) through ultrasound.
* Serum 25-hydroxyvitamin D [25(OH)D] levels below 20 ng/mL (indicating vitamin D deficiency).
* Presence of symptoms associated with uterine fibroid, such as menorrhagia (heavy menstrual bleeding), or bulk-related symptoms (e.g., urinary frequency).
* Participants should be generally healthy, with no history of other chronic illnesses that could affect the study's outcomes (e.g., autoimmune diseases, cancers, severe liver or kidney diseases).
* Willingness to provide written informed consent for participation in the study.
* No current use of hormonal therapy, other vitamin D supplements, or medications known to influence calcium metabolism or uterine fibroid growth (e.g., GnRH agonists, anti-estrogens).
* Participants must be willing and able to adhere to the study protocol, including attending follow-up visits and completing any required assessments or tests.

Exclusion Criteria:

* Women younger than 18 or older than 50 years.
* Serum 25-hydroxyvitamin D [25(OH)D] levels of 20 ng/mL or higher.
* Women without a confirmed diagnosis of uterine fibroids (leiomyoma) through imaging.
* Pregnant or breastfeeding women, or those planning to conceive during the study period.
* Presence of chronic illnesses such as autoimmune diseases, cancers, or severe liver or kidney disease that could interfere with the study's outcomes.
* Current or recent use of hormonal therapy, other vitamin D supplements, or medications that affect calcium metabolism or uterine fibroid growth (e.g., GnRH agonists, anti-estrogens).
* Women who have undergone surgical interventions (e.g., myomectomy, hysterectomy) or other medical treatments specifically for uterine fibroid within the past 6 months.
* Women with conditions like hyperparathyroidism or calcium disorders that might affect vitamin D metabolism or fibroid growth.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Effect of Vitamin D3 supplementation on symptomatic uterine fibroid in women with Vitamin D deficiency. | 18 months
  Fibroid size by cm

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Bangabandhu Sheikh Mujib medical university, Dhaka, Sahabag
  - Bangabandhu Sheikh Mujib medical university, Dhaka

IPD SHARING:
Plan to Share IPD: No